CLINICAL TRIAL: NCT07404475
Title: Relationship Between Microcirculatory Alterations and Coagulopathy in Sepsis: Prospective Observational Study.
Brief Title: Microcirculation and Coagulopathy in Sepsis
Acronym: [MicroCOAG]
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Prof., Università Politecnica delle Marche
Other Study IDs: Micro_COAG_2023
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Coagulopathy
Keywords: sepsis; microcirculation; tissue oxygenation; coagulopathy; glycocalyx
MeSH Terms: conditions — Sepsis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis-induced coagulopathy (SIC) and microvascular dysfunction are hallmark features of sepsis, yet their longitudinal relationship remains poorly understood. The aim of this study is to investigate the interplay between sublingual microcirculation, endothelial damage, peripheral tissue oxygenation and coagulation parameters in patients with sepsis.

DETAILED DESCRIPTION:
Prospective observational study. Inclusion criteria: adult (>18 years of age) patients with sepsis or septic shock. Exclusion criteria:sepsis for more than 24 hours, pre-existing coagulopathy (severe liver disease, inherited bleeding disorders), concurrent use of therapeutic anticoagulation or thrombolytic agents, factors impeding the sublingual microvascular assessment (including maxillo-facial trauma or recent oral surgery) pregnancy and inability to obtain informed consent. For all patients we will record age, gender, admission diagnosis, source of sepsis, comorbidities, the Sequential Organ Failure Assessment (SOFA), the Acute Physiology and Chronic Evaluation II (APACHE II) and the Simplified Acute Physiology Score II (SAPS II). Clinical and laboratory data will be collected daily from day 0 to day 4, including mean arterial pressure (MAP), heart rate (HR), arterial lactate levels, use of sedatives, vasoactive agents with dosage and anticoagulant angents. At day 0, arterial blood samples will be withdrawn and immediately centrifuged; plasma samples will be stored at -70°C for measurement of Syndecan-1 and thrombomodulin levels.Standard coagulation laboratory tests will be analysed daily from day 0 to day 4, including platelet count, international normalized ratio (INR), activated partial thromboplastin time (aPTT), fibrinogen, antithrombin and D-dimer levels. The sepsis-induced coagulopathy (SIC) and the disseminated intravascular coagulation (DIC) scores will be calculated daily. Thromboelastography will be performed daily. The sublingual microcirculation will be assessed on day 0 and day 4 to evaluate parameters of vessel density and microvascular flow quality. Near Infrared Spectroscopy will be used on day 0 to evaluate tissue (thenar eminence) O2 saturation and its dynamic changes during a vascular occlusion test, providing indices of tissue O2 extraction capacity and microvascular reactivity.Data from previous studies suggest that at least 50% of patients with sepsis present with coagulopathy. The hypothesis underlying this study is that patients who develop sepsis-induced coagulopathy exhibit more severe microcirculatory alterations at the time of sepsis diagnosis. In a previous study involving septic patients, we observed a baseline Perfused Vessel Density (PVD) of 22.8±4.7 mm/mm2. Based on these data, and assuming a mean difference in PVD of at least 20% (±5%) between patients who develop SIC and those who do not (unpaired samples t-test), it was calculated that a total sample size of 30 patients would be sufficient to demonstrate a statistically significant difference with a power of 80% and an alpha error of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years of age)
* sepsis or septic shock

Exclusion Criteria:

* sepsis for more than 24 hours
* pre-existing coagulopathy
* concurrent use of therapeutic anticoagulation or thrombolytic agents
* factors impeding the sublingual microvascular assessment
* pregnancy
* inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with sepsis or septic shock admitted to a 14-bed medical Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Perfused vessel density | day 0 (on enrollment)
  difference between patients with sepsis induced coagulopathy and patients without coagulopathy

SECONDARY OUTCOMES:
variations in microvascular parameters | day 0 to day 4 (96 hours)
  evolution of microcirculatory alterations in patients with or without coagulopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria delle Marche, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No